CLINICAL TRIAL: NCT06916247
Title: Evaluation of MA Proactive Care Program Using Cost Prediction Model With Randomized Waitlist
Brief Title: Evaluation of AI Cost Prediction Model to Enroll Patients in Complex Care Management Program
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Richard K. Leuchter, MD, Assistant Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB-24-0849
Record Dates: First submitted 2025-03-21; First posted 2025-04-08 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Chronic Disease
Keywords: High utilization; Complex care management; Cost prediction model
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Complex Care Management (Active Comparator): Patients randomized to be contacted for enrollment into the complex care management program called ProActive Care.
  Interventions: Behavioral: Complex care management program
- Care as usual (No Intervention): Patient randomized to be put on a waitlist for being contacted for enrollment into ProActive Care (ie, not enrolled in ProActive Care).

INTERVENTIONS:
Behavioral: Complex care management program — Intensive outpatient care management program that includes contact from nurses and case managers to help coordinate care, detect clinical red flags, and reduce overall unplanned acute care utilization.
  Arms: Complex Care Management

SUMMARY:
Currently, UCLA Health (specifically the Office of Population Health and Accountable Care, or OPHAC) runs a complex care management program called Proactive Care (goal is to reduce care utilization by providing personalized care navigation/case management). Every month, an AI Population Risk tool runs to identify around 250 of the 480,000 or so UCLA primary care patients, and RNs contact these 250 patients to enroll in Proactive Care. Starting in December 2024, OPHAC launched a new method of enrolling UCLA's Medicare Advantage (MA) patients into Proactive Care: an AI Cost Prediction model. The idea is the same-- the top 250 highest predicted cost patients will be enrolled in Proactive Care. The investigators will evaluate this model and subsequent enrollment into the program by randomizing the waitlist of MA patients waiting to enroll in Proactive Care, thereby creating a control group. The top 500 highest predicted cost patients will be identified each month, and following a 1:1 randomization, 250 will be contacted for enrollment and the rest will be put on a wait-list control group for 10 months unless otherwise requested by their provider to be enrolled in the Proactive Care program earlier.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Enrolled in a UCLA Managed Care Plan
* Cost prediction model identifies patient as having high predicted costs over the next 12 months

Exclusion Criteria:

* Currently enrolled in any UCLA care management program
* Enrolled in any UCLA care management program in the last 12 months
* Already has an active referral to a care management program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2024-08-16 (Actual); Primary Completion 2025-09-09 (Actual); Study Completion 2026-05-12 (Estimated)

PRIMARY OUTCOMES:
Days alive and out of hospital (DAOH) at 120 days from randomization | 120 days after randomization
  The sum of the number of days that a patient is not hospitalized under inpatient or observation status, and alive, out of a maximum of 120 days post-randomization.

SECONDARY OUTCOMES:
Days alive and out of hospital (DAOH) at 30 days from randomization | 30 days after randomization
  The sum of the number of days that a patient is not hospitalized under inpatient or observation status, and alive, out of a maximum of 30 days post-randomization.
Days alive and out of hospital (DAOH) at 90 days from randomization | 90 days after randomization
  The sum of the number of days that a patient is not hospitalized under inpatient or observation status, and alive, out of a maximum of 90 days post-randomization.
Days alive and out of hospital (DAOH) at 10 months from randomization | 10 months post-randomization
  The sum of the number of days that a patient is not hospitalized under inpatient or observation status, and alive, out of a maximum of 300 days post-randomization.
Total healthcare expenditures at 10 months from randomization | 10 months post-randomization
  The sum of all healthcare expenditures (inpatient, outpatient, prescription, etc.) as determined by claims data.
All-cause hospitalizations at 10 months from randomization | 10 months post-randomization
  The total number of hospitalizations under inpatient or observation status for any cause
All-cause emergency department visits at 10 months from randomization | 10 months post-randomization
  The total number of emergency department visits that did not result in hospitalization, for any cause.
All-cause mortality at 10 months from randomization | 10 months post-randomization
  The total number of deaths from any cause
Ambulator contact days | 10 months post-randomization
  The number of days a patient spends outside the home receiving health care, defined as the total number of days with a primary care or specialty care office visit, test, imaging, procedure, or treatment

OTHER OUTCOMES:
Cost prediction model performance over 22 months, as measured by area under the receiver operating characteristic curve | 12 months after the final cohort enrolls
  Observed healthcare expenditures for each month's control cohort will be measured over the subsequent 12 months after randomization (ie, 10 months of enrollment + 12 months of follow-up= 22 months), and compared to model-predicted healthcare expenditures. This analysis will only be conducted in the control group, as the intervention is designed to affect healthcare expenditures in the treatment group.
Protocol fidelity over the 10 months of enrollment | 14 months post-randomization
  The sum of two metrics:
  * The proportion of patients randomized to the intervention who enroll in the complex care management program
  * The proportion of patients randomized to the control who do not enroll in the complex care management program.
Avoidable hospitalizations | 10 months post-randomization
  The number of hospitalizations that could have been avoided through timely access to ambulatory care
Avoidable emergency department visits | 10 months post-randomization
  The number of emergency department visits that could have been avoided through timely access to ambulatory care

CONTACTS AND LOCATIONS:
Overall Officials: Richard K Leuchter, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Health, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-03-31): https://cdn.clinicaltrials.gov/large-docs/47/NCT06916247/SAP_000.pdf